CLINICAL TRIAL: NCT02998411
Title: Population Pharmacokinetics Approaches for the Optimization of Anti-infective Concentrations Among Hospitalized Patients
Brief Title: Population Pharmacokinetics of Anti-infectives in Hospitalized Patients
Acronym: OptiPOP
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI16012
Record Dates: First submitted 2016-11-16; First posted 2016-12-20 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Patient Receiving Anti-infectives Whatever Disease
Keywords: anti-infectives; adults; pharmacokinetic; pharmacodynamic end-points; clinical cure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AI treatment and dosage
  Interventions: Other: Titration

INTERVENTIONS:
Other: Titration

SUMMARY:
In case of sepsis, the therapeutic success is strongly influenced by the choice of anti-infectives (AI) in terms of spectrum, dosage and administration schedule. It is therefore critical to achieve adequate AI concentration as quickly as possible.

This protocol aims to define a common framework to studies conducted jointly by the Antimicrobial Stewardship Tea, the Pharmacology department of Cochin hospital and within the APHP Centre hospital group for various AI in a range of specific study populations (intensive care unit patients, neutropenic patients…).

These studies will use mathematical modeling methodologies to investigate the pharmacokinetics (PK) and pharmacodynamics (PD) of different AI including PK/PD targets or any other biological compartment. The effects of covariates on PK and PD parameters will be investigated to better explain the between-subject variability (BSV) and to ultimately suggest individualized dosage regimens.

DETAILED DESCRIPTION:
Patients with sepsis who receive inadequate AI regimen have a high risk of poor clinical outcomes. It is therefore critical to achieve adequate concentration of the AI as quickly as possible in these patients.

Pharmacokinetics (PK) describes the drug concentration-time courses in body fluids resulting from administration of a certain drug dose, pharmacodynamics (PD) the observed effect resulting from a certain drug concentration. The three PK/PD indices most commonly evaluated for AI are: the ratio of the maximal unbound drug concentration to the MIC (fCmax/MIC), the ratio of the area under the unbound drug concentration-time curve to the MIC (fAUC/MIC) or the percentage of a 24 h time period where the unbound drug concentration exceeds the MIC (fT.MIC). Dosing regimens are chosen to reach a target value of the main PK/PD index.

In hospitalized patients, a high between-subject variability is expected on PK parameters, related to the severity of the disease (sepsis, neutropenia, organ failure...), weight, age (geriatric patients, neonates...) and the co-administration of other medications leading to potential drug interactions. The PD variability is strongly influenced by the immune status, type of infection, inoculum size, comorbidities.

The optiPOP protocol aims to define a common framework to PK/PD studies conducted jointly by the Antimicrobial Stewardship Team, the Pharmacology department of Cochin hospital and within the APHP Centre hospital group.

These studies will use mathematical population pharmacokinetic modeling methodologies to investigate PK/PD parameters of various AI in a range of specific study populations (ICU, neutropenic patients…). The effects of covariates on PK and PD parameters will be investigated in order to better explain the between-subject variability and to ultimately suggest individualized dosage regimens.

OptiPOP is a prospective, non-interventional, single center study, based on data regularly collected during the therapeutic drug monitoring of AI.

The antimicrobial stewardship team (AST) has a role in advising clinicians for the diagnostic and treatment of infectious diseases. It is closely involved in daily therapeutic drug monitoring of AI, in collaboration with the department of pharmacology and within the APHP Centre hospital group. Patient selection will take place in all medical and surgical wards of the hospital. The AST senior physician will check the eligibility criteria and propose the study to the patient, in accordance with the referring physician. Any adult patient requiring the administration of an AI with at least one plasma concentration measurement or any other biological compartment conducted in Cochin department of pharmacology and within the APHP Centre hospital group will be eligible. The AST physician will give a briefing note to the patient, and the non-oral opposition for the retrieval and analysis of data will be collected.

No intervention or no charge will be made for this study. It is planned to include 60 patients per molecule.

ELIGIBILITY:
Inclusion Criteria:

* Every adult hospitalized in Cochin hospital, receiving an AI and who require at least one AI concentration measurement or any other biological compartment in the Cochin department of pharmacology

Exclusion Criteria:

* Patient having notified to the physician the refusal for data recovery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients hospitalized in Cochin hospital receiving an AI agent and who require at least one AI concentration measurement or any other biological compartment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Anti-infectives concentration | 28 days

SECONDARY OUTCOMES:
Composite measure of the health condition | 28 days
  Clinical and laboratory data : anthropometric characteristics; organs function, severity score, type of infection, micro-organsim and sensitivity, infectious biological parameters
Minimum Inhibitory Concentration (MIC) of the suspected or documented pathogen | 28 days
  Pharmacodynamic characteristics of the molecule

CONTACTS AND LOCATIONS:
Overall Officials: Etienne CANOUI, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin Hospital, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No